CLINICAL TRIAL: NCT05868395
Title: Efficacy of Polatuzumab, Bendamustine and Rituximab in Patients With Relapsed/ Refractory Mantle Cell Lymphoma - a Single Center Phase II Trial
Brief Title: Efficacy of Polatuzumab, Bendamustine and Rituximab in Patients With Relapsed/ Refractory Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Kiesewetter, Ap. Prof. Priv.-Doz. DDr, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Polatuzumab-BR in r/r MCL
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Mantle-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — polatuzumab vedotin; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polatuzumab, bendamustine and rituximab (Experimental): Polatuzumab vedotin 1.8 mg/kg i.v. on day 2 of cycle 1, then on day 1 of each subsequent cycle, bendamustine 90 mg/m2 i.v. day 2 & 3 of cycle 1, then on day 1 & 2 of each subsequent cycle and rituximab 375 mg/m2 i.v. on day 1 of each cycle every 3 weeks.
  Interventions: Drug: Polatuzumab, bendamustin und rituximab

INTERVENTIONS:
Drug: Polatuzumab, bendamustin und rituximab — * Polatuzumab vedotin 1.8 mg/kg i.v. on day 2 of cycle 1, then on day 1 of each subsequent cycle
  * Bendamustine 90 mg/m2 i.v. day 2 & 3 of cycle 1, then on day 1 & 2 of each subsequent cycle
  * Rituximab 375 mg/m2 i.v. on day 1 of each cycle
  * Each cycle is 21 days long
  * Up to 6 cycles per patients planned
  Other Names: Polivy; Bendamustin; Mabthera

SUMMARY:
Polatuzumab, bendamustine and rituximab in patients with relapsed/ refractory mantle cell lymphoma

DETAILED DESCRIPTION:
Polatuzumab vedotin will be administered at a dose of 1.8 mg/kg i.v. on day 2 of cycle 1, then on day 1 of each subsequent cycle.

Bendamustine will be administered at a dose 90 mg/m2 i.v. day 2 & 3 of cycle 1, then on day 1 & 2 of each subsequent cycle.

Rituximab will be administered at a dose 375 mg/m2 i.v. on day 1 of each cycle. Each cycle is 21 days long Response rate by RECIST 1.1 is definied as the primary study endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Capability of understanding the purpose of the study and have given written informed consent.
* Age greater than or equal to 18 years
* Histologically or cytologically confirmed relapsed or refractory MCL
* r/r MCL patients following standard first line chemotherapy who have received at least one prior regimen including ibrutinib
* If the participant has received prior bendamustine, response duration must have been > 1 year
* Presence of at least one lymph node or mass measurable for response
* Life expectancy of at least 24 weeks
* ECOG 0-2
* Adequate hematological, renal and hepatic function unless inadequate function is due to underlying disease

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (MAbs or recombinant antibody-related fusion proteins) or known sensitivity or allergy to bendamustine or rituximab
* Contraindications to polatuzumab, bendamustine or rituximab
* Prior use of any MAb, radioimmunoconjugate, or antibody-drug conjugate (ADC) within 4 weeks or 5 half-lives before cycle 1 day 1
* Use of any investigational agent within 28 days prior to initiation of study treatment
* History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 3 years
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to cycle 1 day
* Major surgery or significant traumatic injury within 28 days of the first dose of study drug
* Ongoing corticosteroid use >30 mg per day prednisone or equivalent, for purposes other than lymphoma symptom control
* Autologous stem cell transplant (SCT) within 100 days prior to cycle 1 day 1
* Prior allogeneic SCT
* Eligibility for autologous SCT
* Primary or secondary CNS lymphoma
* Current grade >1 peripheral neuropathy
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks prior to Cycle 1 Day 1
* Suspected or latent tuberculosis
* Positive test results for chronic hepatitis B virus (HBV) infection or for hepatitis C virus (HCV) antibody
* Known history of human immunodeficiency virus (HIV) seropositive status or known infection with human T-cell leukemia virus 1 (HTLV-1) virus
* Women who are pregnant or lactating or who intend to become pregnant within a year of the last dose of study treatment. Women of childbearing potential must have a negative pregnancy test at screening, pregnancy testing must be performed within 7 days before first administration of IMP. Approved methods of birth control must be used
* Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to the last dose of protocol therapy. Adequate contraception defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.
* Male subjects unable or unwilling to use adequate contraception methods.
* Evidence of laboratory abnormalities in standard renal, hepatic, or coagulation function tests

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2027-05-24 (Estimated); Study Completion 2027-05-24 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From date of enrollment until the date of first documented progression or date of death from any cause or treatmentdiscontinuation from any other reason, whichever came first, assessedup to 36 months]
  Objective response rate according to RECIST 1.1

SECONDARY OUTCOMES:
Survival | From date of inclusion until the date of first documented progression or date of death from any cause or treatmentdiscontinuation from any other reason, whichever came first, assessedup to 36 months]
  Progression-free survival (PFS), Event-free survival (EFS), Overall survival (OS)
Safety / Toxicity | From date of inclusion until the date of first documented progression or date of death from any cause or treatmentdiscontinuation from any other reason, whichever came first, assessedup to 36 months]
  Safety / Toxicity according to Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Kiesewetter, MD, Principal Investigator — Medical University Vienna
Locations (1):
- AKH Vienna, Division of Oncology Department of Medicine I, Vienna, Austria